CLINICAL TRIAL: NCT04117048
Title: Evaluation of the Impact of Using LabPad® Point-of-care to Measure International Normalized Ratio (INR) at Home on the Patient's Follow up on VKA
Brief Title: INR at Home Measurement by the LabPad® Point-of-care in Patients on Vitamin K Antagonist Drugs (VKA)
Acronym: INRADOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medicalps (Other)
Collaborators: AG2R La Mondiale (Other); AVALUN (Unknown); Icadom (Industry); ORIADE NOVIALE (Unknown); SIL-LAB INNOVATIONS (Unknown); TASDA (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RCB 2019-A01357-50
Record Dates: First submitted 2019-10-03; First posted 2019-10-07 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-02

CONDITIONS: Vitamine K Antagonist (VKA) Treatment; International Normalized Ratio (INR) Measure at Home; Thromboembolic Pathology
Keywords: INR; Labpad®; VKA

STUDY DESIGN:
Intervention Model Description: All patients included benefit from at home INR measure
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- At home INR measurement with LabPad® (Experimental): All at home INR measurements will be performed with the LabPad® point-of-care
  Interventions: Device: LabPad® point-of-care

INTERVENTIONS:
Device: LabPad® point-of-care — All at home INR measurements will be performed by the nurse using the LabPad® point-of-care

SUMMARY:
This study evaluates the impact of using LabPad® point-of-care to measure International Normalized Ratio (INR) at home on the patient's follow up on vitamine K antagonist (VKA) treatment during 6 months.

DETAILED DESCRIPTION:
The impact of the LabPad® point-of-care use by the nurse will be evaluated in the patients on vitamine K antagonist (VKA) treatment by measuring the time elapsed between the reading of the International Normalized Ratio (INR) by the LabPad® at patient's home and the validation of the biological measure, The time that the patient spends in his therapeutic range will be measured. The adverse events related to VKA will also be collected. At the end of the study, the patient will complete satisfaction and usage questionnaires about the LabPad®.

This study will be performed for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age
* Patient treated with VKA and without any heparin - VKA relay
* Patient able to read and understand the procedure, and able to express consent for the study

Exclusion Criteria:

* Patient treated with heparin
* Patient treated with direct oral anticoagulants (DAOs)
* Patient with antiphospholipid antibody syndrome (APA)
* Patient not available or wishing to change region within one year of inclusion
* Patient currently participating or having participated in the month preceding the inclusion in another interventional clinical research that may impact the study, this impact is left to the investigator's discretion
* Persons referred to in Articles L.1121-5 to L.1121-8 of the French Public Health Law (corresponds to all protected persons: pregnant woman (verified by the dosage of β- human chorionic gonadotropin for any woman wishing to participate in the protocol and of childbearing age < 60 years), parturient, nursing woman, person deprived of liberty by judicial or administrative decision, person subject to a legal protection measure)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2019-10-03 (Actual); Primary Completion 2020-04-03 (Actual); Study Completion 2020-04-03 (Actual)

PRIMARY OUTCOMES:
Patient follow up time, regardless of the value of the INR | During 6 months of use
  Measure of time in minute elapsed between the reading of the INR by the LabPad® and the validation of the biological measure, regardless of the value of the INR

SECONDARY OUTCOMES:
Patient follow up time, in case of INR outside the safety interval (≤1,8 or ≥5) | During 6 months of use
  Measure of time in minute elapsed between the reading of the INR by the LabPad® and the validation of the biological measure, in case of INR outside the safety interval (≤1,8 or ≥5)
Time in Therapeutic Range | During 6 months of use
  Measure of the time in hour that patient spends in his therapeutic range
Number of adverse events related to VKA | During 6 months of use
  Collection of adverse events during patient follow-up
Patient's satisfaction about the LabPad®: Satisfaction Questionnaire | After 6 months of use
  The patient will complete a Satisfaction Questionnaire at the end of the study. This is a questionnaire made by ourselves of 9 questions with 7 submissions and the total score will be into a value ranging from the worst satisfaction 7 to the best satisfaction 63.
LabPad® patient's use | After 6 months of use
  The patient will complete a Questionnaire on the LabPad® use at the end of the study.
  This is a scale from 0 (no use desire) to 10 (best use desire) and demographic questions to characterise the patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratoire ORIADE NOVIALE, Saint-Marcellin, France

IPD SHARING:
Plan to Share IPD: No